CLINICAL TRIAL: NCT00771823
Title: A Placebo Controlled Study of the Impact on Insulin Sensitivity and Lipid Profile of Maraviroc 300 mg Twice Daily in HIV Negative Male Volunteers
Brief Title: Maraviroc 300 mg Twice Daily in HIV Negative Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Graeme Moyle, St Stephen's AIDS Trust
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SSAT025; 2007-004477-25 (EudraCT Number)
Record Dates: First submitted 2008-07-28; First posted 2008-10-15 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator)
  Interventions: Drug: Maraviroc
- 1 (Active Comparator): * Maraviroc 300 mg twice daily for the first 14 days of the study.
  * Placebo twice daily for the last 14 days of the study
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc 300 mg twice daily for the first 14 days of the study. Placebo twice daily for the last 14 days of the study
  Arms: 1
Drug: Maraviroc — * Placebo twice daily for the first 14 days of the study.
  * Maraviroc 300 mg twice daily for the last 14 days of the study.
  Arms: 2

SUMMARY:
A placebo controlled study of the impact on insulin sensitivity and lipid profile of maraviroc 300 mg twice daily in HIV negative male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have documented negative HIV serology by ELISA and P24 antigen
* Subjects must be clinically well males aged between 18 to 60 years.
* Fasting blood glucose, total cholesterol and triglycerides within normal limits
* Hepatic transaminases (AST and ALT) ≤ 3 × upper limit of normal (ULN)
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm3; platelets ≥ 50,000/mm3; hemoglobin ≥ 8.0 g/dL)
* Serum amylase ≤ 1.5 × ULN
* Sexually active males must use condoms during the course of the study
* Life expectancy ≥ 1 year
* Willing and able to provide informed consent

Exclusion Criteria:

* Subjects with a waist hip ratio > 0.97 or BMI > 28 kg/m2 will be excluded
* Acute or chronic hepatitis B infection (determined by positive hepatitis B surface antigen result at the screening visit)
* Acute or chronic hepatitis C infection (determined by positive hepatitis C antibody result at the screening visit)
* Other metabolic syndrome or disease process in the opinion of the investigator likely to cause marked disturbance in glucose and lipid homeostasis including hypertension.
* Receiving on-going therapy with any of the following:

  * Metabolically active medications
  * Any lipid-lowering medication
  * Hormonal agents (oestrogens or androgens)
  * Glucocorticoids
  * Beta-blockers
  * Thiazide diuretics
  * Thyroid preparations
  * Psychotropic agents
  * Anabolic steroids
  * Megestrol acetate

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity by euglycaemic clamp method | two weeks

SECONDARY OUTCOMES:
Change from baseline in serum levels of fasting cholesterol, triglycerides Changes in serum biomarkers of vascular inflammation and in CD36 PMBC and other related markers gene expression | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Moyle, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- Chelsea and Westminster Hospital, London, London, United Kingdom